CLINICAL TRIAL: NCT02008539
Title: Treatment of Advanced Gastrointestinal Cancer in a Phase I/II Trial With Modified Autologous MSC_apceth_101
Acronym: TREAT-ME 1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment terminated after 13 patients (14 planned); further patients did not meet eligibility criteria to receive autologous IMP
Sponsor: Apceth GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC_apceth_101/1
Record Dates: First submitted 2013-10-28; First posted 2013-12-11 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Advanced Gastrointestinal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: MSC_apceth_101

INTERVENTIONS:
Drug: MSC_apceth_101

SUMMARY:
To evaluate the safety and tolerability of MSC_apceth_101.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or recurrent or metastatic gastrointestinal adenocarcinoma.
* Premature or scheduled termination of standard therapy
* Progressive disease as clinically assessed by the investigator
* Max. tumour lesion ≤ 5 cm
* Adequate organ function
* Ability of patient to understand character and individual consequences of clinical trial
* Age ≥ 18 years
* Written informed consent must be available before any study specific procedure is performed

Exclusion Criteria:

* Patients with severe heart diseases
* Clinical significant ischemic disease during the last 4 weeks before Visit 1
* Severe lung disease
* Symptomatic peritoneal carcinomatosis
* Symptomatic pleural or pericardial effusion
* Serious uncontrolled acute infections less than 3 weeks before Visit 1
* Known dependency on alcohol or other drugs
* Patients requiring corticoids in doses above the Cushing threshold
* Known liver fibrosis or liver cirrhosis
* Any concomitant severe disease which could compromise the objectives of this study in the judgment of the investigator
* Female patient who is pregnant or breast feeding
* Participation in another clinical trial or observation period, respectively, during the last 4 weeks prior to the first IMP dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as indicated by Common Toxicity Criteria (CTC-AE) of the National Cancer Institute | day 56 (+/- 7) in patient group 1 and day 29 (+/-3) in patient group 2

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Munich, Munich, Germany